CLINICAL TRIAL: NCT05274737
Title: Randomized Trial Comparing A Novel Sling With A Traditional Abduction Sling After Shoulder Surgery
Brief Title: Comparison Of A Novel Sling With A Traditional Abduction Sling After Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orthopedic Institute, Sioux Falls, SD (Other)
Responsible Party: Principal Investigator, Keith Baumgarten, Principal Investigator, Orthopedic Institute, Sioux Falls, SD
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Sling study
Record Dates: First submitted 2022-02-28; First posted 2022-03-10 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Rotator Cuff Tears; Osteo Arthritis Shoulders
Keywords: Shoulder; Sling
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, controlled model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial Immobilization with the novel sling (Experimental): 20 patients will be placed in the novel sling after surgery for the first two weeks. For the second two weeks (days 15-28) they will crossover and utilize the standard abduction sling. For the final two weeks (days 29-42) they will choose their preferred sling type and use it for the remainder of six week immobilization period.
  Interventions: Device: Novel sling
- Initial Postoperative Immobilization with the standard abduction sling (Experimental): 20 patients will be placed in the traditional abduction sling after surgery for the first two weeks. For the second two weeks (days 15-28) they will crossover and utilize the novel sling. For the final two weeks (days 29-42) they will choose their preferred sling type and use it for the remainder of six week immobilization period.
  Interventions: Device: Traditional abduction sling

INTERVENTIONS:
Device: Novel sling — The novel sling was designed and created by the principal investigator to address these concerns of the traditional slings that are currently available for postsurgical protection and immobilization after shoulder surgery. It is anticipated that the novel sling will allow the patient to be more active and more comfortable while still providing a safe healing environment after a shoulder injury or shoulder surgery.
  Arms: Initial Immobilization with the novel sling
Device: Traditional abduction sling — An abduction sling is the most common type of sling utilized to protect patients after rotator cuff surgery and total shoulder of arthroplasty and can be considered the current standard of care.
  Arms: Initial Postoperative Immobilization with the standard abduction sling

SUMMARY:
The objective of this study is to determine if the novel shoulder sling has higher patient satisfaction compared to a traditional, abduction sling with at least equivalent postoperative outcomes after arthroscopic rotator cuff repair and total shoulder arthroplasty.

DETAILED DESCRIPTION:
Specific Aim I:

To determine if patients undergoing arthroscopic rotator cuff repair prefer the traditional abduction sling vs the novel sling.

Specific Aim II:

To determine if patients undergoing total shoulder arthroplasty prefer the traditional abduction sling vs the novel sling.

Specific Aim III:

To determine if short term follow-up (2, 4, 6 weeks), subjective patient-reported outcomes are superior in patients utilizing the novel sling compared to patients utilizing the traditional, abduction sling.

Specific Aim IV:

To determine if longer term follow-up (6 weeks, 14 weeks, 6 months, and 12 months), validated patient-reported outcomes are similar (non-inferior) in patients utilizing the novel sling compared to a historical control cohort of patients that only utilized the traditional, abduction sling. The purpose of this aim is to ensure that patients that utilize the novel novel sling for 2 to 4 weeks (with the traditional sling used for the rest of the 6 week period) do not have inferior outcomes compared to patients that have worn the traditional sling for a total of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroscopic rotator cuff repair and anatomic total shoulder arthroplasty
* Dominant extremity undergoing surgery

Exclusion Criteria:

* Patients undergoing revision surgery
* Patients with a history of significant cervical spine disease, peripheral neuropathy, or concomitant wrist or elbow disorders
* Patients that do not understand English
* Patients unwilling to participate or follow up for the study protocols

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Patient choice of type of sling to utilize from postoperative days 29-42 | 6 weeks after surgery
  Categorical variable of which sling they preferred to use for the last two weeks of their 6 week postoperative immobilization period
Sling satisfaction survey | Prior to surgery
  a novel, sling satisfaction score (SSS)[scale 0= best to 10=worst] utilizing a number-based visual analog scale will be utilized to assess baseline characteristics of common symptoms that have been attributed to sling use
Sling satisfaction survey | 14 days after surgery
  a novel, sling satisfaction score (SSS) [scale 0= best to 10=worst] utilizing a number-based visual analog scale will be utilized to assess baseline characteristics of common symptoms that have been attributed to sling use and satisfaction with the type of sling utilized during this time period
Sling satisfaction survey | 15 days after surgery
  a novel, sling satisfaction score (SSS) [scale 0= best to 10=worst] utilizing a number-based visual analog scale will be utilized to assess baseline characteristics of common symptoms that have been attributed to sling use and satisfaction with the type of sling utilized during this time point. The rationale for recording both the day 14 and day 15 SSS is to get the patient's immediate impression on the potential subjective differences between the slings within 24 hours of changing to the alternate sling.
Sling satisfaction survey | 28 days after surgery
  a novel, sling satisfaction score (SSS) [scale 0= best to 10=worst]utilizing a number-based visual analog scale will be utilized to assess baseline characteristics of common symptoms that have been attributed to sling use and satisfaction with the type of sling utilized during this time period
Sling satisfaction survey | 6 weeks after surgery
  a novel, sling satisfaction score (SSS) [scale 0= best to 10=worst] utilizing a number-based visual analog scale will be utilized to assess baseline characteristics of common symptoms that have been attributed to sling use and satisfaction with the type of sling utilized during this time period
Sling satisfaction survey | 14 weeks after surgery
  a novel, sling satisfaction score (SSS) [scale 0= best to 10=worst] utilizing a number-based visual analog scale will be utilized to assess baseline characteristics of common symptoms that have been attributed to sling use
Sling satisfaction survey | 6 months after surgery
  a novel, sling satisfaction score (SSS) [scale 0= best to 10=worst] utilizing a number-based visual analog scale will be utilized to assess baseline characteristics of common symptoms that have been attributed to sling use
Sling satisfaction survey | 12 months after surgery
  a novel, sling satisfaction score (SSS) [scale 0= best to 10=worst] utilizing a number-based visual analog scale will be utilized to assess baseline characteristics of common symptoms that have been attributed to sling use

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Score | Prior to surgery
  A validated joint specific patient-determined outcome score (low 0 - 100 high)
American Shoulder and Elbow Surgeons Score | 14 weeks after surgery
  A validated joint specific patient-determined outcome score (low 0 - 100 high)
American Shoulder and Elbow Surgeons Score | 6 months after surgery
  A validated joint specific patient-determined outcome score (low 0 - 100 high)
American Shoulder and Elbow Surgeons Score | 12 months after surgery
  A validated joint specific patient-determined outcome score (low 0 - 100 high)
Single Assessment Numeric Evaluation | Prior to surgery
  A validated general patient-determined outcome score (low 0 - 100 high)
Single Assessment Numeric Evaluation | 6 weeks after surgery
  A validated general patient-determined outcome score (low 0 - 100 high)
Single Assessment Numeric Evaluation | 14 weeks after surgery
  A validated general patient-determined outcome score (low 0 - 100 high)
Single Assessment Numeric Evaluation | 6 months after surgery
  A validated general patient-determined outcome score (low 0 - 100 high)
Single Assessment Numeric Evaluation | 12 months after surgery
  A validated general patient-determined outcome score (low 0 - 100 high)
Shoulder Activity Level | Prior to surgery
  A validated shoulder-specific activity score (low 0 - 20 high)
Shoulder Activity Level | 14 weeks after surgery
  A validated shoulder-specific activity score (low 0 - 20 high)
Shoulder Activity Level | 6 months after surgery
  A validated shoulder-specific activity score (low 0 - 20 high)
Shoulder Activity Level | 12 months after surgery
  A validated shoulder-specific activity score (low 0 - 20 high)

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Institute, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is not a plan to allow IPD with other researchers